CLINICAL TRIAL: NCT03645954
Title: Femoral Triangle and Adductor Canal Blocks Versus Femoral Nerve Block for Total Knee Arthroplasty: Postoperative Pain Management and Functional Recovery
Brief Title: Femoral Triangle and Adductor Canal Blocks Versus Femoral Nerve Block for Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lithuanian University of Health Sciences (Other)
Responsible Party: Principal Investigator, Inna Jaremko, Principal Investigator, Lithuanian University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BEC-MF-172
Record Dates: First submitted 2018-08-15; First posted 2018-08-24 (Actual); Results first posted 2021-01-13 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-01

CONDITIONS: Total Knee Arthroplasty
Keywords: Femoral triangle block; Adductor canal block; Femoral nerve block; Primary total knee arthroplasty; Pain management; Functional recovery
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Femoral Nerve Block (Active Comparator): The femoral nerve block will be performed under the ultrasound guidance by a single injection of local anesthetic around all the femoral nerve branches inside the proximal part of the femoral triangle.
  Interventions: Procedure: Femoral Nerve Block
- Femoral Triangle & Adductor Canal Blocks (Active Comparator): These two blocks will be performed together.
  Firstly, the femoral triangle block will be performed under the ultrasound guidance by a single injection of local anesthetic at the level where the medial border of the sartorius muscle intersects the medial border of the adductor longus muscle. Local anesthetic will be injected laterally to the femoral artery.
  Secondly, the adductor canal block will be performed under the ultrasound guidance by a single injection of local anesthetic at the level where the femoral vessels (artery and vein) dive deeper from the sartorius muscle. Local anesthetic will be injected under the femoral artery.
  Interventions: Procedure: Femoral Triangle & Adductor Canal Blocks

INTERVENTIONS:
Procedure: Femoral Nerve Block — Procedure: Femoral Nerve Block
  The femoral nerve block will be performed as described in Arms section.
  Device: Ultrasound
  Linear ultrasound transducer probe (Flex Focus 400 exp, bk medical, Denmark) will be used to guide the needle placement.
  Device: Needle
  20-gauge 50 mm Ultraplex needle (B. Braun Medical Inc., Melsungen, Germany) will be used to perform the femoral nerve block.
  Drug: Local anesthetic
  Bupivacaine 0.125% 20 mL will be used to perform the femoral nerve block.
  Arms: Femoral Nerve Block
Procedure: Femoral Triangle & Adductor Canal Blocks — Procedure: Femoral Triangle & Adductor Canal Blocks
  These two blocks will be performed as described in Arms section.
  Device: Ultrasound
  Linear ultrasound transducer probe (Flex Focus 400 exp, bk medical, Denmark) will be used to guide the needle placement.
  Device: Needle
  20-gauge 100 mm Ultraplex needle (B. Braun Medical Inc., Melsungen, Germany) will be used to perform the femoral triangle block and adductor canal block.
  Drug: Local anesthetic
  Bupivacaine 0.125% 20 mL will be used to perform the femoral triangle block and adductor canal block (10 mL for each block).
  Arms: Femoral Triangle & Adductor Canal Blocks

SUMMARY:
This prospective, double-blinded, randomized controlled study evaluates effects of femoral triangle and adductor canal blocks in comparison with femoral nerve block for primary total knee arthroplasty. Patients undergoing primary total knee arthroplasty will be randomly assigned to receive either femoral triangle and adductor canal blocks or femoral nerve block. Comparison of these two groups of patients will be based on the effects on postoperative pain control, extent of motor blockade, ability of early ambulation, patients satisfaction rates over the time of clinical recovery and the length of hospitalization.

To the investigator's knowledge, no comparison has been made between femoral triangle and adductor canal blocks and femoral nerve block or any other block. Consequently, we hypothesized that femoral triangle and adductor canal blocks and femoral nerve block provide similar effects on postoperative pain control, but femoral triangle and adductor canal blocks are superior to femoral nerve block in terms of early postoperative mobilization.

DETAILED DESCRIPTION:
The aim: to evaluate femoral triangle and adductor canal blocks and femoral nerve block regarding the postoperative analgesic efficacy, extent of motor blockade, ability of early ambulation in patients following primary total knee arthroplasty.

Primary Hypothesis: femoral triangle and adductor canal blocks and femoral nerve block provide similar postoperative pain relieving effect after primary total knee arthroplasty.

Secondary Effects: femoral triangle and adductor canal blocks provide better ability of early ambulation after primary total knee arthroplasty.

The objectives:

1. To compare postoperative pain control effects between femoral triangle and adductor canal blocks and femoral nerve block groups of patients after primary total knee joint replacement surgery.
2. To assess the ability of early ambulation and extent of motor blockade after primary total knee joint replacement surgery between the groups of patients.
3. To estimate opioid consumption and its adverse effects in femoral triangle and adductor canal blocks and femoral nerve block groups of patients after primary total knee arthroplasty.
4. To compare patients postoperative satisfaction rates between femoral triangle and adductor canal blocks and femoral nerve block groups of patients after primary total knee arthroplasty.

Methods:

The prospective, double-blinded study includes American Society of Anesthesiologists (ASA) physical status I-III in preoperative assessment, aged 18-90 years, admitted for primary total knee arthroplasty. Preoperatively patients will be blindly randomized into one of two groups: femoral triangle and adductor canal blocks group and femoral nerve block group. Group assignment will be concealed by opaque envelopes that will be opened only after the enrollment. The anesthesiologist performing the block will be aware of the treatment, but the participant and outcomes assessor will be blinded to the group assignment.

All blocks will be performed by the anesthesiologist under the guidance of a linear ultrasound transducer probe. Femoral nerve block will be performed at the proximal part of the femoral triangle by 20 mL of 0.125% bupivacaine injection. Femoral triangle and adductor canal blocks will be performed together. Femoral triangle block will be performed at the level where the medial border of the sartorius muscle intersects the medial border of the adductor longus muscle with injection of 10 mL of 0.125% bupivacaine. Local anesthetic will be injected laterally to the femoral artery. Adductor canal block will be performed at the level where the femoral vessels (artery and vein) dive deeper from the sartorius muscle with injection of 10 mL of 0.125% bupivacaine. Local anesthetic will be injected under the femoral artery.

During the perioperative period all patients from both groups will receive a standardized anesthetic and analgesic. Premedication of midazolam 2.5-5 mg and dexamethasone 4 mg will be given to all patients and a slow fluid infusion of crystalloids with 1 g of tranexamic acid and 10 mg of ketamine will be started once as an intravenous cannula will be placed. Spinal anesthesia after identification of the subarachnoid space will be performed with 15 mg of levobupivacaine. After that, femoral triangle and adductor canal blocks or femoral nerve block (depending on the group of patients) will be performed under the ultrasound guidance. Patients will be sedated with intravenously administered propofol during the surgery. The local infiltration analgesia will be performed by the surgeon at the end of surgery with combination of 30 mL of 0.5% bupivacaine, 0.3 mL of 0.1% adrenaline and 90 mL of 0.9% sodium chloride. After the surgery patients will be transferred to the post-anesthesia care unit (PACU).

During the postoperative period for analgesia NSAIDs will be available to both groups of patients. NSAIDs such as dexketoprofen 50 mg will be administered 2 times and acetaminophen 1 g will be administered 3 times per day. Opioids will also be available to patients as intramuscular boluses of pethidine 50 mg or morphine 10 mg without restriction and administered for moderate or severe pain (VAS pain score of 5 or greater out of 10).

Postoperative pain control efficacy will be assessed at 3, 6, 24 and 48 hours after surgery using visual analogue scale (VAS) from 0 to 10 (0 - no pain, 10 - worst imaginable pain) at rest, during active and passive 45 degree knee flexion. The requirement of additional analgesics and their adverse effects (if any) will be recorded.

The extent of motor blockade will be evaluated at 3, 6, 24, 48 hours after surgery. Patients will be asked to flex the foot, to flex the knee and to lift up the straight leg. The possible leg motion at 3, 6, 24 and 48 hours postoperatively will be assessed with Bromage scale grades: Grade I - free movement of legs and feet, Grade II - just able to flex knees with free movement of feet, Grade III - unable to flex knees, but with free movement of feet, Grade IV - unable to move legs or feet.

Patients ability of early ambulation will be evaluated using Timed Up and Go (TUG) test at 24 and 48 hours after surgery. To do the TUG test, patients will have to sit down on the bed, get up from the bed, walk 3 meters forward, turn, walk back 3 meters to the bed and sit down. The time taken by a patient to perform this test will be calculated with a chronometer.

After the conversation with each patient and assessment of postoperative pain control efficacy, extent of motor blockade, ability of early ambulation, the rate of patient satisfaction will be evaluated using a 10 point scale from 0 (completely unsatisfied) to 10 (totally satisfied) at 3, 6, 24, 48 hours after surgery.

The length of hospital stay and rate of complications (if any), including falls, local anesthetic toxicity or neurological complications, will be recorded in both groups of patients.

According to study protocol, both groups of patients will be compared in terms of postoperative pain control, opioid consumption, extent of motor blockade, ability of early ambulation, patients satisfaction rates over the time of clinical recovery and the length of hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing primary unilateral total knee arthroplasty under the spinal anesthesia.
* Age 18 - 90 years.
* Patients conformed to American Society of Anesthesiologists (ASA) physical status I-III in preoperative assessment.
* Ability to follow the study protocol.

Exclusion Criteria:

* Inability or refusal to follow the study protocol.
* American Society of Anesthesiologists (ASA) physical status classification of IV or higher.
* Coagulopathy.
* Pre-existing lower extremity neuromuscular disorders.
* Local infection over the injection site.
* Allergy or contraindications to the drugs used in the study (local anesthetics, NSAIDs, opioids).
* Chronic opioid use.
* Other type of anesthesia.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2018-08-28 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arunas Gelmanas, MDPhDAssProf, Study Chair — Lithuanian University of Health Sciences
Locations (1):
- Lithuanian University of Health Sciences Kauno Klinikos, Department of Anesthesiology, Kaunas, Lithuania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bendtsen TF, Moriggl B, Chan V, Borglum J. The Optimal Analgesic Block for Total Knee Arthroplasty. Reg Anesth Pain Med. 2016 Nov/Dec;41(6):711-719. doi: 10.1097/AAP.0000000000000485. PMID 27685346
- [Background] Kuang MJ, Ma JX, Fu L, He WW, Zhao J, Ma XL. Is Adductor Canal Block Better Than Femoral Nerve Block in Primary Total Knee Arthroplasty? A GRADE Analysis of the Evidence Through a Systematic Review and Meta-Analysis. J Arthroplasty. 2017 Oct;32(10):3238-3248.e3. doi: 10.1016/j.arth.2017.05.015. Epub 2017 May 17. PMID 28606458
- [Background] Grevstad U, Mathiesen O, Lind T, Dahl JB. Effect of adductor canal block on pain in patients with severe pain after total knee arthroplasty: a randomized study with individual patient analysis. Br J Anaesth. 2014 May;112(5):912-9. doi: 10.1093/bja/aet441. Epub 2014 Jan 8. PMID 24401802
- [Background] Seo SS, Kim OG, Seo JH, Kim DH, Kim YG, Park BY. Comparison of the Effect of Continuous Femoral Nerve Block and Adductor Canal Block after Primary Total Knee Arthroplasty. Clin Orthop Surg. 2017 Sep;9(3):303-309. doi: 10.4055/cios.2017.9.3.303. Epub 2017 Aug 4. PMID 28861197
- [Background] Koh IJ, Choi YJ, Kim MS, Koh HJ, Kang MS, In Y. Femoral Nerve Block versus Adductor Canal Block for Analgesia after Total Knee Arthroplasty. Knee Surg Relat Res. 2017 Jun 1;29(2):87-95. doi: 10.5792/ksrr.16.039. PMID 28545172
- [Background] Dong CC, Dong SL, He FC. Comparison of Adductor Canal Block and Femoral Nerve Block for Postoperative Pain in Total Knee Arthroplasty: A Systematic Review and Meta-analysis. Medicine (Baltimore). 2016 Mar;95(12):e2983. doi: 10.1097/MD.0000000000002983. PMID 27015172

RESULTS

PARTICIPANT FLOW:
Groups:
- Femoral Nerve Block: The femoral nerve block was performed under the ultrasound guidance by a single injection of Bupivacaine 0.125% 20 mL around all the femoral nerve branches inside the proximal part of the femoral triangle.
- Femoral Triangle & Adductor Canal Blocks: These two blocks will be performed together. The femoral triangle block will be performed under the ultrasound guidance by a single injection of Bupivacaine 0.125% 10 mL at the level where the medial border of the sartorius muscle intersects the medial border of the adductor longus muscle. Local anesthetic will be injected laterally to the femoral artery. The adductor canal block will be performed under the ultrasound guidance by a single injection of Bupivacaine 0.125% 10 mL at the level where the femoral artery and vein dive deeper from the sartorius muscle. Local anesthetic will be injected under the femoral artery.
Period: Overall Study
Arm/Group | Femoral Nerve Block | Femoral Triangle & Adductor Canal Blocks
Started | 40 | 40
Completed | 37 | 40
Not Completed | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Femoral Nerve Block | Femoral Triangle & Adductor Canal Blocks | Total
Number analyzed (Participants) | 37 | 40 | 77
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.1 (9.3) | 68.5 (9.8) | 68.8 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 11 | 35
  Male | 13 | 29 | 42
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 31.9 (5.5) | 31.2 (5.7) | 31.5 (5.6)
Physical Status According to ASA [Count of Participants; unit: Participants] — ASA I - a normal healthy patient ASA II - a patient with mild systemic disease ASA III - a patient with severe systemic disease ASA IV - a patient with severe systemic disease that is a constant threat to life ASA V - a moribund patient who is not expected to survive without the operation ASA VI - a declared brain-dead patient whose organs are being removed for donor purposes
  Participants
    ASA status: I | 2 | 2 | 4
    ASA status: II | 33 | 36 | 69
    ASA status III | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Extent of Motor Blockade
Description: The extent of postoperative motor blockade will be evaluated using Bromage scale: Grade I - free movement of legs and feet, Grade II - just able to flex knees with free movement of feet, Grade III - unable to flex knees, but with free movement of feet, Grade IV - unable to move legs or feet. It will be assessed at 3, 6, 24, 48 hours after surgery.
Time Frame: 3, 6, 24, 48 hours after primary total knee arthroplasty.
Measure: Count of Participants; unit: Participants
Arm/Group | Femoral Nerve Block | Femoral Triangle & Adductor Canal Blocks
Number analyzed (Participants) | 37 | 40
Participants
  3 hours after TKA: Bromage Grade I | 18 | 29
  3 hours after TKA: Bromage Grade II | 13 | 5
  3 hours after TKA: Bromage Grade III | 1 | 1
  3 hours after TKA: Bromage Grade IV | 5 | 5
  6 hours after TKA: Bromage Grade I | 25 | 38
  6 hours after TKA: Bromage Grade II | 12 | 2
  6 hours after TKA: Bromage Grade III | 0 | 0
  6 hours after TKA: Bromage Grade IV | 0 | 0
  24 hours after TKA: Bromage Grade I | 31 | 35
  24 hours after TKA: Bromage Grade II | 6 | 5
  24 hours after TKA: Bromage Grade III | 0 | 0
  24 hours after TKA: Bromage Grade IV | 0 | 0
  48 hours after TKA: Bromage Grade I | 29 | 34
  48 hours after TKA: Bromage Grade II | 8 | 6
  48 hours after TKA: Bromage Grade III | 0 | 0
  48 hours after TKA: Bromage Grade IV | 0 | 0
Statistical Analysis 1: Comparison: Femoral Nerve Block vs Femoral Triangle & Adductor Canal Blocks; Test type: Superiority; p < 0.01, Chi-squared — The threshold for statistical significance was p = 0.05

2. Primary Outcome: Postoperative Pain Intensity and Pain Control
Description: Postoperative pain intensity and pain control will be assessed in both groups using visual analogue scale (VAS). VAS scale is consisted of a scale from 0 (no pain) to 10 (worst imaginable pain). Pain control and pain intensity will be assessed at rest, during active and passive 45 degree knee flexion at 3, 6, 24, 48 hours after surgery.
Time Frame: 3, 6, 24, 48 hours after primary total knee arthroplasty.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Femoral Nerve Block | Femoral Triangle & Adductor Canal Blocks
Number analyzed (Participants) | 37 | 40
score on a scale
  3 hours after TKA (at rest) | 1.22 (2.04) | 0.45 (1.11)
  6 hours after TKA (at rest) | 1.27 (1.97) | 1.45 (2.06)
  24 hours after TKA (at rest) | 2.00 (2.24) | 2.10 (2.13)
  48 hours after TKA (at rest) | 1.78 (2.45) | 1.63 (1.81)
  3 hours after TKA (passive 45-degree knee flexion) | 2.14 (2.76) | 1.10 (1.89)
  6 hours after TKA (passive 45-degree knee flexion) | 2.27 (2.32) | 2.55 (2.40)
  24 hours after TKA (passive 45-degree knee flexion) | 4.41 (2.39) | 3.73 (2.24)
  48 hours after TKA (passive 45-degree knee flexion) | 4.19 (2.61) | 3.40 (2.01)
  3 hours after TKA (active 45-degree knee flexion) | 2.19 (2.81) | 1.20 (1.93)
  6 hours after TKA (active 45-degree knee flexion) | 2.35 (2.40) | 2.63 (2.53)
  24 hours after TKA (active 45-degree knee flexion) | 5.00 (2.63) | 4.33 (2.43)
  48 hours after TKA (active 45-degree knee flexion) | 4.54 (2.65) | 3.95 (2.24)
Statistical Analysis 1: Comparison: Femoral Nerve Block vs Femoral Triangle & Adductor Canal Blocks; Test type: Superiority; p > 0.05, t-test, 2 sided — The threshold for statistical significance was p = 0.05

3. Secondary Outcome: Ability of Early Ambulation After Surgery
Description: Postoperative ability of early ambulation will be assessed using Timed Up and Go (TUG) test. The TUG test measures the time it takes the patient to get up from a bed, walk 3 meters, turn, walk back to the bed and sit down. The TUG test results will be evaluated at 24 and 48 hours after surgery.
Time Frame: 24, 48 hours after primary total knee arthroplasty.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Femoral Nerve Block | Femoral Triangle & Adductor Canal Blocks
Number analyzed (Participants) | 37 | 40
seconds
  24 hours after TKA | 53.6 (54.8) | 53.7 (23.0)
  48 hours after TKA | 47.3 (47.1) | 36.9 (15.2)
Statistical Analysis 1: Comparison: Femoral Nerve Block vs Femoral Triangle & Adductor Canal Blocks; Test type: Other; p > 0.05, t-test, 2 sided — The threshold for statistical significance was p = 0.05

4. Secondary Outcome: Number of Participants Needing Additional Opioids
Description: The need of additional opioids will be recorded at 3, 6, 24 and 48 hours after surgery in both groups.
Time Frame: 3, 6, 24, 48 hours after primary total knee arthroplasty.
Measure: Count of Participants; unit: Participants
Arm/Group | Femoral Nerve Block | Femoral Triangle & Adductor Canal Blocks
Number analyzed (Participants) | 37 | 40
Participants
  3 hours after TKA | 5 | 3
  6 hours after TKA | 8 | 13
  24 hours after TKA | 27 | 23
  48 hours after TKA | 24 | 22
Statistical Analysis 1: Comparison: Femoral Nerve Block vs Femoral Triangle & Adductor Canal Blocks; Test type: Other; p > 0.05, Chi-squared — The threshold for statistical significance was p = 0.05

5. Secondary Outcome: Rate of Patients Satisfaction
Description: Patient satisfaction rates will be evaluated using a 10 point scale from 0 (completely unsatisfied) to 10 (totally satisfied) at 3, 6, 24, 48 hours after surgery.
Time Frame: 3, 6, 24, 48 hours after primary total knee arthroplasty.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Femoral Nerve Block | Femoral Triangle & Adductor Canal Blocks
Number analyzed (Participants) | 37 | 40
score on a scale
  3 hours after TKA | 8.8 (1.4) | 8.9 (1.8)
  6 hours after TKA | 8.5 (1.5) | 8.8 (1.7)
  24 hours after TKA | 8.1 (1.7) | 8.4 (1.5)
  48 hours after TKA | 8.1 (1.8) | 8.6 (1.3)
Statistical Analysis 1: Comparison: Femoral Nerve Block vs Femoral Triangle & Adductor Canal Blocks; Test type: Other; p > 0.05, t-test, 2 sided — The threshold for statistical significance was p = 0.05

6. Secondary Outcome: Number of Participants With Nausea or Vomiting
Description: The number of patients with nausea and vomiting will be evaluated in both groups of patients.
Time Frame: 3, 6, 24, 48 hours after primary total knee arthroplasty.
Measure: Count of Participants; unit: Participants
Arm/Group | Femoral Nerve Block | Femoral Triangle & Adductor Canal Blocks
Number analyzed (Participants) | 37 | 40
Participants
  3 hours after TKA: Nausea | 1 | 1
  3 hours after TKA: Vomiting | 0 | 0
  3 hours after TKA: No nausea or vomiting | 36 | 39
  6 hours after TKA: Nausea | 2 | 1
  6 hours after TKA: Vomiting | 0 | 1
  6 hours after TKA: No nausea or vomiting | 35 | 38
  24 hours after TKA: Nausea | 3 | 3
  24 hours after TKA: Vomiting | 0 | 1
  24 hours after TKA: No nausea or vomiting | 34 | 36
  48 hours after TKA: Nausea | 1 | 1
  48 hours after TKA: Vomiting | 1 | 0
  48 hours after TKA: No nausea or vomiting | 35 | 39
Statistical Analysis 1: Comparison: Femoral Nerve Block vs Femoral Triangle & Adductor Canal Blocks; Test type: Other; p > 0.05, Chi-squared — The threshold for statistical significance was p = 0.05

ADVERSE EVENTS:
Time Frame: 3, 6, 24, 48 hours after surgery
Description: All-Cause Mortality was not monitored/assessed.
Groups:
- Femoral Nerve Block: The femoral nerve block will be performed under the ultrasound guidance by a single injection of local anesthetic around all the femoral nerve branches inside the proximal part of the femoral triangle.
  Femoral Nerve Block: Procedure: Femoral Nerve Block
  The femoral nerve block will be performed as described in Arms section.
  Device: Ultrasound
  Linear ultrasound transducer probe (Flex Focus 400 exp, bk medical, Denmark) will be used to guide the needle placement.
  Device: Needle
  20-gauge 50 mm Ultraplex needle (B. Braun Medical Inc., Melsungen, Germany) will be used to perform the femoral nerve block.
  Drug: Local anesthetic
  Bupivacaine 0.125% 20 mL will be used to perform the femoral nerve block.
- Femoral Triangle & Adductor Canal Blocks: These two blocks will be performed together.
  Firstly, the femoral triangle block will be performed under the ultrasound guidance by a single injection of local anesthetic at the level where the medial border of the sartorius muscle intersects the medial border of the adductor longus muscle. Local anesthetic will be injected laterally to the femoral artery.
  Secondly, the adductor canal block will be performed under the ultrasound guidance by a single injection of local anesthetic at the level where the femoral vessels (artery and vein) dive deeper from the sartorius muscle. Local anesthetic will be injected under the femoral artery.
  Femoral Triangle & Adductor Canal Blocks: Procedure: Femoral Triangle & Adductor Canal Blocks
  These two blocks will be performed as described in Arms section.
  Device: Ultrasound
  Linear ultrasound transducer probe (Flex Focus 400 exp, bk medical, Denmark) will be used to guide the needle placement.
  Device: Needle
  20-gauge 100 mm Ultraplex needle (B. Braun Medical Inc., Melsungen, Germany) will be used to perform the femoral triangle block and adductor canal block.
  Drug: Local anesthetic
  Bupivacaine 0.125% 20 mL will be used to perform the femoral triangle block and adductor canal block (10 mL for each block).
Arm/Group | Femoral Nerve Block | Femoral Triangle & Adductor Canal Blocks
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/40
Other Adverse Events (participants affected / at risk) | 0/37 | 0/40

LIMITATIONS AND CAVEATS:
There is no control group of patients who would not receive any peripheral nerve block.

We were not able to measure the quadriceps muscle strenght with a dynamometer.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-24): https://cdn.clinicaltrials.gov/large-docs/54/NCT03645954/Prot_SAP_001.pdf